CLINICAL TRIAL: NCT03808207
Title: Human Milk Lipid Profile Assessment and Influences of Mother's Diet Valutazione Del Profilo Lipidico Del Latte Materno e Della Sua Variazione in Relazione Alla Dieta Materna
Brief Title: Human Milk Lipid Profile Assessment and Influences of Mother's Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Fanaro Silvia, Assistant Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HM2018
Record Dates: First submitted 2018-10-01; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Breastfeeding; Human Milk; Diet Habit; Fatty Acid; Infant Growth
Keywords: Docosahexaenoic acid; LcPufas; Diet; Human milk; gas chromatography
MeSH Terms: conditions — Breast Feeding; Feeding Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Blind randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The lipid profile will be assessed by an external investigator who is blind for the dietary advices and choices of the single patient. Milk samples are assigned a progressive numerical code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Increase of the average intake of dietary DHA: dietary advices concerning the concentration of docosahexaenoic acid (DHA) in several foods; the recommended daily or weekly intake of different food options (animal, vegetal) in order to reach the average intake of 300-350 mg DHA/day
  Interventions: Other: Dietary counseling and DHA dietary increase in breastfeeding mothers
- Control group (No Intervention): No specific dietary advice; Only endorsement and promotion of breastfeeding.

INTERVENTIONS:
Other: Dietary counseling and DHA dietary increase in breastfeeding mothers — Specific dietary advices in order to increase the daily/weekly intake of docosahexaenoic acid of breastfeeding mothers for the first 3 months after delivery
  Arms: Intervention group

SUMMARY:
Human milk profile is unique and diet exerts a pivot role in determing its composition.

As a rule, nursing mothers do not receive specific nutritional indications aimed at improving the lipid profile of milk, despite the scientific evidence in favor of the importance of DHA in the infant's diet.

The research aims to determine the effect of a dietary counseling specifically targeted at increasing the intake of fatty acids ω3 (DHA, EPA and ALA) on the lipid profile of breast milk, in order to identify effective and viable nutrition claims for breastfeeding women.

DETAILED DESCRIPTION:
Breast milk, with its unique and inimitable characteristics, is the ideal feeding for full-term babies. The maternal diet strongly influences the composition of milk, in particular, its lipid proflie, which provides about 50% of the infant's energy needs. In particular, the polyunsaturated fatty acid fraction may varies according ethnic origin and diet habit.

Docosahexaenoic acid or DHA (22: 6 n-3), a long chain fatty acid from the omega 3 series, plays a fundamental role in neurogenesis and neurotransmission as well as in vision, as it is present in both brain, particularly in neural synapses, and in retinal photoreceptors. In particular, the brain grows rapidly from birth to the first year of life, and this growth must be supported by the adequate and balanced intake of all fatty acids; among these we have seen that DHA has a priority role. Observational studies have shown that higher concentrations in breast milk and / or maternal and / or neonatal DHA blood are associated with greater visual acuity, language development, psychomotor development, attention and higher IQ scores in children. The paucity of DHA in the maternal diet of Western countries, and the low conversion rate of α-linolenic acid or ALA (18: 3 n-3) in DHA in humans babies, may result in an insufficient supply for the newborn brain.

Most of the prospective studies carried out in this area have evaluated the effects of maternal supplementation of fish oils, algal oils, chia oil, linseed oil. At present, the positive association between the frequency of fish consumption and DHA levels in breast milk has only been evaluated in retrospective studies.

On these basis, the purpose of this randomized clinical trial is the evaluation of the efficacy of a dietary counseling specifically aimed at increasing the intake of ALA and its long-chain derivatives on the lipid profile of breast milk. Women in the intervention group will be provided an informative scheme on food options with the highest content of the aforementioned polyunsaturated fatty acids. The expected result, at 3 months after delivery, in the intervention group is an increase of DHA in breast milk 80% higher than the value found in the control group (women on a free diet). Dietary habits at enrollment and actual intakes will be recorded for 1 week before the two milk samplings. The research is also aimed at verifying the efficacy of a nutritional educational intervention, without strict preordained schemes, and above all without the aid of dietary supplements.

ELIGIBILITY:
Inclusion Criteria:

* women who have delivered at > 33 weeks GA
* ongoing breastfeeding
* consent received

Exclusion Criteria:

* contraindications to breastfeeding
* neonatal malformations or genetic anomalies
* language barrier

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — mother's milk; breastfeeding status
Enrollment: 24 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Human milk lipid profile assesment after 3 months of DHA/ALA diet enrichment | 80 days
  Lipid profile assesment of human milk at 10 days and 3 months after delivery. Evaluation of the effect of DHA/ALA diet enrichment during the study period. Measurement of total fat (g/100 ml), saturated fatty acids, monounsaturated fatty and polyunsaturated fatty acids concentration (mg/100 ml), and specifically LA, ALA, ARA, DHA and EPA concentration (mg/100 ml) will be performed with gas chromatograph coupled to a MS / MS mass spectrometer.

SECONDARY OUTCOMES:
Lipid profile characteristics in human milk of mothers delivering preterm or term infants | 80 days
  Lipid profile characteristics in human milk of mothers who delivered 34-36 weeks and 6 days or >37 weeks gestational age infants.
  Measurement of total fat (g/100 ml), saturated fatty acids, monounsaturated fatty and polyunsaturated fatty acids concentration (mg/100 ml), and specifically LA, ALA, ARA, DHA and EPA concentration (mg/100 ml) will be performed with gas chromatograph coupled to a MS / MS mass spectrometer.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Fanaro, MD, Principal Investigator — Medical Science Department, University of Ferrara, Italy
Locations (1):
- UO Neonatal Intensive Care Unit and Neonatology, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03808207/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03808207/ICF_001.pdf